CLINICAL TRIAL: NCT04173676
Title: Sentinel Lymph Node Navigation Using Near-infrared Imaging in Radical Esophagectomy Surgery ：a Single-arm Clinical Trial
Brief Title: Sentinel Lymph Node Navigation Surgery Using Near-infrared Imaging in Early Esophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: No.ZDWY[2018]LunziNo.(K31-1)
Record Dates: First submitted 2019-11-17; First posted 2019-11-22 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-05

CONDITIONS: Detection Rate of SLN ; Accuracy Rate of Lymph Node Metastasis
MeSH Terms: interventions — Indocyanine Green; Injections

STUDY DESIGN:
Intervention Model Description: The sentinel lymph nodes are observed by submucosal injection of ICG
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of indocyanine green (Experimental): submucosal injection of ICG is by gastroscopy on the superior and inferior edge of the esophageal tumor,Dose of 0.5mg
  Interventions: Drug: Indocyanine Green for Injection

INTERVENTIONS:
Drug: Indocyanine Green for Injection — The sentinel lymph nodes were observed by submucosal injection of ICG

SUMMARY:
The esophageal squamous cell carcinoma (ESCC) has high prevalence and mortality in China, which become a severe challenge for public health. Esophagectomy is the preferred choice for the patients who are diagnosed with ESCC in early stage .Although three-field lymphadenectomy has improved patient survival and reduced tumor recurrence, Surgery-related complications increased dramatically.

It has become a research hotspot to find an effective detection method to identify the lymph node metastasis of ESCC and avoid ineffective expanded lymphadenectomy .The molecular imaging technology has been developed for intra-operative visualization and precise resection of the tumors.

Indocyanine Green for Injection (ICG) has been used as a contrast agent in the near-infrared imaging system for the surgical navigation technology, which has a relatively positive effect in the clinical application of gastric cancer and liver cancer.There are few reports on the application of ICG near-infrared imaging tracer lymph nodes in the surgery of ESCC. This study intends to identify the detection rate of sentinel lymph node (SLN) and determine the accuracy of regional lymph node metastasis in ESCC by ICG near-infrared imaging technique, which provides clinical evidence for subsequent precise resection of the lymph nodes.

This will be one-arm prospective trial. The ESCC patients will be recruited with strict criteria. 84 patients will be enrolled between18 and 75 years old, without gender limit. The submucosal injection of ICG will be performed preoperatively by gastroscopy on the superior and inferior edge of the esophageal tumor. NIR fluorescence imaging will be performed intraoperatively to observe the lymph nodes. The luminescent lymph node is defined as SLN. According to the standard procedure, 3 field lymphadenectomy will be performed, and all the resected lymph nodes will be subjected to pathological analysis including correlation study of fluorescence signal and tumor tissue in pathology slice.

This clinical trial is anticipated to evaluate the detection rate of SLN in ESCC with ICG near-infrared fluorescence imaging and determine the accuracy of regional lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old, gender is not limited;
2. patient who is diagnosed with ESCC and choose to proceed with surgery
3. patient with cTNM stage:T1-3N0-1M0
4. tumor located at the middle thoracic or lower thoracic esophagus
5. The main organ function is basically normal: Karnofsky score >70%;
6. Laboratory blood tests meet surgical standards;

Exclusion Criteria:

1. pregnancy or breastfeeding
2. history of iodide or seafood allergy,
3. Patient with occult metastatic disease at the time of surgery
4. patient with mental disorder;
5. Patient who is simultaneously involved in another clinical trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
the detection rate of sentinel lymph node | through study completion, an average of 1 year
  the detection rate of sentinel lymph node in all the enrolled patients
The positive rate of sentinel lymph node | through study completion, an average of 1 year
  the positive rate of sentinel lymph node in all the enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shirakawa S, Toyama H, Kido M, Fukumoto T. A prospective single-center protocol for using near-infrared fluorescence imaging with indocyanine green during staging laparoscopy to detect small metastasis from pancreatic cancer. BMC Surg. 2019 Nov 7;19(1):165. doi: 10.1186/s12893-019-0635-0. PMID 31699083
- [Result] Lim HJ, Chiow AKH, Lee LS, Tan SS, Goh BK, Koh YX, Chan CY, Lee SY. Novel method of intraoperative liver tumour localisation with indocyanine green and near-infrared imaging. Singapore Med J. 2021 Apr;62(4):182-189. doi: 10.11622/smedj.2019137. Epub 2019 Nov 4. PMID 31680180
- [Result] Yanagi Y, Yoshimaru K, Matsuura T, Shibui Y, Kohashi K, Takahashi Y, Obata S, Sozaki R, Izaki T, Taguchi T. The outcome of real-time evaluation of biliary flow using near-infrared fluorescence cholangiography with Indocyanine green in biliary atresia surgery. J Pediatr Surg. 2019 Dec;54(12):2574-2578. doi: 10.1016/j.jpedsurg.2019.08.029. Epub 2019 Sep 2. PMID 31575415
- [Result] Hayami S, Matsuda K, Iwamoto H, Ueno M, Kawai M, Hirono S, Okada K, Miyazawa M, Tamura K, Mitani Y, Kitahata Y, Mizumoto Y, Yamaue H. Visualization and quantification of anastomotic perfusion in colorectal surgery using near-infrared fluorescence. Tech Coloproctol. 2019 Oct;23(10):973-980. doi: 10.1007/s10151-019-02089-5. Epub 2019 Sep 18. PMID 31535238
- [Result] Zhou SC, Tian YT, Wang XW, Zhao CD, Ma S, Jiang J, Li EN, Zhou HT, Liu Q, Liang JW, Zhou ZX, Wang XS. Application of indocyanine green-enhanced near-infrared fluorescence-guided imaging in laparoscopic lateral pelvic lymph node dissection for middle-low rectal cancer. World J Gastroenterol. 2019 Aug 21;25(31):4502-4511. doi: 10.3748/wjg.v25.i31.4502. PMID 31496628
- [Result] Yamada Y, Ohno M, Fujino A, Kanamori Y, Irie R, Yoshioka T, Miyazaki O, Uchida H, Fukuda A, Sakamoto S, Kasahara M, Matsumoto K, Fuchimoto Y, Hoshino K, Kuroda T, Hishiki T. Fluorescence-Guided Surgery for Hepatoblastoma with Indocyanine Green. Cancers (Basel). 2019 Aug 20;11(8):1215. doi: 10.3390/cancers11081215. PMID 31434361
- [Result] Predina JD, Newton AD, Corbett C, Shin M, Sulfyok LF, Okusanya OT, Delikatny EJ, Nie S, Gaughan C, Jarrar D, Pechet T, Kucharczuk JC, Singhal S. Near-infrared intraoperative imaging for minimally invasive pulmonary metastasectomy for sarcomas. J Thorac Cardiovasc Surg. 2019 May;157(5):2061-2069. doi: 10.1016/j.jtcvs.2018.10.169. Epub 2018 Dec 14. PMID 31288365
- [Result] Pennathur A, Gibson MK, Jobe BA, Luketich JD. Oesophageal carcinoma. Lancet. 2013 Feb 2;381(9864):400-12. doi: 10.1016/S0140-6736(12)60643-6. PMID 23374478
- [Result] Rice TW, Apperson-Hansen C, DiPaola LM, Semple ME, Lerut TE, Orringer MB, Chen LQ, Hofstetter WL, Smithers BM, Rusch VW, Wijnhoven BP, Chen KN, Davies AR, D'Journo XB, Kesler KA, Luketich JD, Ferguson MK, Rasanen JV, van Hillegersberg R, Fang W, Durand L, Allum WH, Cecconello I, Cerfolio RJ, Pera M, Griffin SM, Burger R, Liu JF, Allen MS, Law S, Watson TJ, Darling GE, Scott WJ, Duranceau A, Denlinger CE, Schipper PH, Ishwaran H, Blackstone EH. Worldwide Esophageal Cancer Collaboration: clinical staging data. Dis Esophagus. 2016 Oct;29(7):707-714. doi: 10.1111/dote.12493. PMID 27731549
- [Result] Lerut T, Nafteux P, Moons J, Coosemans W, Decker G, De Leyn P, Van Raemdonck D, Ectors N. Three-field lymphadenectomy for carcinoma of the esophagus and gastroesophageal junction in 174 R0 resections: impact on staging, disease-free survival, and outcome: a plea for adaptation of TNM classification in upper-half esophageal carcinoma. Ann Surg. 2004 Dec;240(6):962-72; discussion 972-4. doi: 10.1097/01.sla.0000145925.70409.d7. PMID 15570202
- [Result] Taniyama Y, Nakamura T, Mitamura A, Teshima J, Katsura K, Abe S, Nakano T, Kamei T, Miyata G, Ouchi N. A strategy for supraclavicular lymph node dissection using recurrent laryngeal nerve lymph node status in thoracic esophageal squamous cell carcinoma. Ann Thorac Surg. 2013 Jun;95(6):1930-7. doi: 10.1016/j.athoracsur.2013.03.069. Epub 2013 May 1. PMID 23642437
- [Derived] Wang X, Hu Y, Wu X, Liang M, Hu Z, Gan X, Li D, Cao Q, Shan H. Near-infrared fluorescence imaging-guided lymphatic mapping in thoracic esophageal cancer surgery. Surg Endosc. 2022 Jun;36(6):3994-4003. doi: 10.1007/s00464-021-08720-7. Epub 2021 Sep 7. PMID 34494149